CLINICAL TRIAL: NCT06171776
Title: Evaluation of Conservative Management of Teeth With Deep Cavitated Carious Lesions Using Three Different Lining Materials-a Randomized Clinical Trial
Brief Title: Evaluation of Conservative Management of Teeth With Deep Cavitated Carious Lesions
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Magdy Moustafa, Lecturer of esthetic and conservative dentistry, faculty of dentistry, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 345
Record Dates: First submitted 2023-11-29; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Deep Caries; Pulp Exposure, Dental
MeSH Terms: conditions — Dental Pulp Exposure | interventions — mineral trioxide aggregate; Pemetrexed; TheraCal; fuji IX

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- fuji XI (Active Comparator): chemically cured glass ionomer
  Interventions: Drug: Fuji IX
- RetroMTA (Experimental): cacium silicat cement
  Interventions: Drug: RetroMTA
- Theracal LC (Experimental): resin based calcium silicate cement
  Interventions: Drug: TheraCal

INTERVENTIONS:
Drug: RetroMTA — calcium silicate lining material work as dentin substitute
  Other Names: MTA
  Arms: RetroMTA
Drug: TheraCal — calcium silicat material light cured
  Other Names: resin based calcium silicat
  Arms: Theracal LC
Drug: Fuji IX — filling material bonded chemically to the tooth structure
  Other Names: chemically cured glass
  Arms: fuji XI

SUMMARY:
The goal of this clinical trial is to compare postoperative pain of calcium silicate cement and resin-based tricalcium silicate (TheraCal LC) versus chemically Cured Glass Ionomer cement (FujiXI) in conservative management of very deep carious lesions by selective caries removal

DETAILED DESCRIPTION:
p-Patients having Permanent posterior teeth with very deep carious lesions I 1 calcium silicate cement I 2= resin-based tricalcium silicate (TheraCal LC) C- chemically Glass Ionomer cement O- Outcome name Measuring Device Measuring Unit Primary1ry postoperative pain 1- Refrigerant spray (endo frost ) 2- Percussion (Marchi et al. 2006) 3- Palpation Binary Secondry2ry Peri-apical pathosis Digital radiograph (Hashem et al. 2015) Binary

T- one month, three months, six months,12 months,24 months evaluation S-Randomized clinical trial 7- Trial design: Randomized Controlled Trial. Trial type: single blind parallel arms design Trial framework: Equivalence frame, Allocation ratio: 1:1. Research question In patients having permanent posterior teeth with very deep carious lesions will calcium silicate cement or resin-based tricalcium silicate (TheraCal LC) in comparison to chemically cured glass ionomer cement result in clinical and radiographical success? Methods: Participants, interventions, and outcomes 8-Study Settings: This clinical trial will be held in the Faculty of Oral & Dental Medicine Cairo University, Egypt.

9- Eligibility criteria:

1. Eligibility Criteria of participants:

   Inclusion Criteria of participants:
   1. Patients male or female older than 18 y in good general health
   2. A minimum of 1 deep carious lesion penetrating three-quarters or more into the dentine as identified with the periapical (PA) radiograph; Clinically according to International Caries Detection and Assessment System (ICDAS II) score 4
   3. Clinical symptoms of reversible pulpitis
   4. Positive pulp response to electric pulp test or thermal stimulation
   5. No PA changes viewed on PA radiograph

   Exclusion Criteria of participants:
   1. Clinical symptoms of irreversible pulpitis requiring endodontic treatment
   2. Presence of fistulas or swelling
   3. Mobile teeth or tenderness to percussion
   4. Anterior teeth with aesthetic concerns
   5. Pregnant women, in view of requirements for radiographs
   6. Patients younger than 18 y
   7. Patients unable to give consent
2. Exclusion criteria of the teeth:

   Teeth with symptoms of irreversible pulpitis including persistent dull throbbing pain, sharp spontaneous pain, or pain exacerbated by lying down will be excluded. In addition, patients will be withdrawn from the study if pulp exposure occurred during the baseline operative intervention.
3. Assessor and Operator criteria:

   Operator: O.M. (PHD), Assessor: A.R. (PHD) 10a- Interventions: • Pre-operative clinical assessment :
   1. Thermal testing using Refrigerant spray (Endo Frost, Roeko, Langenau, Germany)
   2. percussion test
   3. Palpation and clinical examination for the signs of inflammation (pain, abscess, sinus tract, and mobility).
   4. PA radiographs using digital radiograph will be taken at baseline (T0) and will be assessed to exclude any signs of irreversible pulpitis (widening of periodontal ligament [PDL] or PA lesions).

      These tests were carried out at baseline, pre-operatively, and at 1 month , 3, 6,12 and 24-month in post-operative follow-up visits
      * Caries removal procedure:

      Local anesthesia will be given to the patient then complete isolation to the tooth using rubber dame the operator O.M. will open the enamel if needed using high speed hand piece (NSK, NSK America Corp,USA) with high speed diamond round bur (Standard shank Ø1.6mm x 19mm FG. Diamond medium grit) (komet Rock Hill, SC, United States) under copious irrigation. Then in caries removal from the walls carbon-steel rose-head bur (komet Rock Hill, SC, United States) in low speed hand piece (W&H DentalwerkBürmoos GmbH, Bürmoos, Austria).Finally the deeper caries will be removed using spoon excavator (no 49, 61 or 73, Dentsply,Maillefer) leaving the last layer affected dentine without any direct pulp exposure (Clarkson et al., 2021) Intervention: RetroMTA (BioMTA, Seoul, Korea) and TheraCal LC (Bisco Inc., Schaumburg, IL, USA) *The material will be applied according to manufacturer instructions

      Comparator: GC Fuji IX GP® (GC America Inc, Alsip, IL,USA) *The material will be applied according to manufacturer instructions Final restoration application: Filtek™ Z250 Universal Restorative (3M Canada, London, Ontario Canada)

      Adhesive system:

      Scotchbond Universal Etchant (3M ESPE, St. Paul MN, USA) & Single Bond Universal adhesive (3M ESPE, St. Paul MN, USA).

      * The material will be applied according to manufacturer instruction as follows: Etchant will be applied for 15 seconds then rinsed for 15 seconds, then cavity will be dried using gentle air stream. Adhesive material will be applied to the cavity and rubbed for 20 second, then will be air thinned using gentle air for 5 seconds and photo-cured for 20 seconds using LED light curing unit. After applying the adhesive, composite will be applied then photo-cured for 40 seconds using LED light curing unit.

   11b-Restoration will be removed when there are any signs of leakage, fracture or sever postoperative pain due to pulpal response and will unergo endodontic treatment.

   13- Radiographical assessment: digital periapical radiograph ( FONA XDC , FONA SRL, Assago, Italy ) will be tacken by A.R. at T0 (after the operative procedure) and after 1 month(T1), 3 (T3) ,6 ( T6) , 12( T12) and 24 ( T24) months using paralleling technique to standardize the final record for each patient then processed in ( DIGORA optime, sordexTuusula, Finland) .

   11- Outcomes: outcomes criteria, measuring devices, scores, characteristics, measuring unite: Criterion M. device Score Characteristics M. unit

   13- Recruitment: Patients will be recruited byA.R. from clinic of conservative dentistry department in Faculty of Oral &Dental Medicine Cairo University, where there is a continuous and high patient flow from which eligible patients will be recruited to fulfill the eligibility criteria 1 week before intervention.

   Methods: Assignment of interventions

   Allocation:

   15a- Sequence generation: Simple randomization will be done by generating numbers from 1:99 using Random Sequence Generator, Randomness and Integrity Services Ltd (https://www.random.org/) .

   No from 1-33 represents the first intervention and from 34-66 is second intervention and from 67-99 is the comparator.

   15b- Allocation concealment: Operator O.M. will choose between numbers in an opaque sealed envelope, which will be arranged by A.R. who will not be involved in any of the phases of the clinical trial. The side to which intervention or control is assigned will be recorded on a computer by O.M. and all records of all patients will be kept with A.R 16- Blinding: The operator will not be blinded to material assignment because of the difference in the application protocol of the restorative materials, which prohibited blinding of the operator; however, assessors will be blinded to the material assignment.

   Methods: Data collection, management, and analysis 17a- Data collection methods:
   * Baseline data collection:

   For every patient medical and dental history will be taken. Examination charts will be filled by A.R

ELIGIBILITY:
Inclusion Criteria:

1. Patients male or female older than 18 y in good general health
2. A minimum of 1 deep carious lesion penetrating three-quarters or more into the dentine as identified with the periapical (PA) radiograph; 3-Clinically according to International Caries Detection and Assessment System (ICDAS II) score 4 (Clinical symptoms of reversible pulpitis)

4. Positive pulp response to thermal stimulation (cold test) 5. No PA changes viewed on PA radiograph

Exclusion Criteria:

1-Clinical symptoms of irreversible pulpitis requiring endodontic treatment 2. Presence of fistulas or swelling 3. Mobile teeth or tenderness to percussion 4. Anterior teeth with aesthetic concerns 5. Pregnant women, in view of requirements for radiographs 6. Patients younger than 18 y 7. Patients unable to give consent

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain (binary) | one week to 24 months
  pain after restoration of teeth using cold test

SECONDARY OUTCOMES:
periapical pathosis detection using digital periapical radiograph | one week to 24 months
  detection of periapical pathosis

CONTACTS AND LOCATIONS:
Locations (1):
- Omnia Magdy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No